CLINICAL TRIAL: NCT03976089
Title: Promoting Healthy Development With the Recipe 4 Success Intervention: A Randomized Controlled Trial
Brief Title: Promoting Healthy Development With the Recipe 4 Success Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Penn State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Recipe4Success
Record Dates: First submitted 2019-06-03; First posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Obesity; Poverty
MeSH Terms: conditions — Obesity | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: 2-arm randomized controlled trial comparing new home visit intervention delivered within Early Head Start to treatment as usual Early Head Start
Who Masked: Outcomes Assessor
Masking Description: Families were randomly assigned to condition and either started new Recipe 4 Success home visits for 10 weeks or continued the standard Early Head Start home visits they had been receiving. Interviewers collecting all outcome data were blind to study condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recipe 4 Success intervention (Experimental): 10 lessons delivered across 10 successive weeks within Early Head Start infrastructure by families' regular Early Head Start home visitors. Lessons involved active coaching in which parents and children prepared healthy snacks or meals. Lessons also included information on children's self-regulation skills and healthy eating habits.
  Interventions: Behavioral: Recipe 4 Success
- Treatment as usual Early Head Start (Active Comparator): Regular Early Head Start home visitors continued to implement evidence-informed developmentally appropriate curriculum designed to promote children's physical health, cognitive skills, and social-emotional functioning as well as parents' capacities to support their children's development.
  Interventions: Behavioral: Treatment as Usual Early Head Start

INTERVENTIONS:
Behavioral: Recipe 4 Success — The Recipe 4 Success intervention consisted of 10 weekly lessons in which parents and toddlers prepared simple snacks or meals.
  All Recipe 4 Success lessons started and ended with some evidence-based information for the parents about children's self-regulation skills or healthy eating habits. Most of each lesson in Recipe 4 Success was devoted to the snack or meal preparation activities. Each week, home visitors coached the parents as they worked with their toddlers to make increasingly challenging snacks and meals. During these activities, home visitors pointed out opportunities for parents to practice sensitive scaffolding strategies. At the same time, these meal and snack preparation activities allowed children to practice multiple age-appropriate self-regulation skills.
  Arms: Recipe 4 Success intervention
Behavioral: Treatment as Usual Early Head Start — Treatment as Usual Early Head Start consisted of an evidence-based curriculum (usually Parents as Teachers) in which home visitors and parents worked with children on activities to support their physical, cognitive, and social-emotional development.
  Arms: Treatment as usual Early Head Start

SUMMARY:
10-session home visit intervention conducted within Early Head Start and designed to reduce low-income toddler's obesity risk and improve their self-regulation skills and parents' sensitivity.

DETAILED DESCRIPTION:
Recipe 4 Success, the product of a university-community engagement collaboration, uses 10 tightly sequenced, structured, and scripted food preparation lessons, delivered as part of Early Head Start home visits, to help low-income parents learn to sensitively scaffold their toddler's self-regulation skills and establish more healthy eating habits. The intervention relies on an active coaching therapeutic approach to deliver content. Recipe 4 Success is focused on parents because their feeding practices influence children's diet, and interventions to prevent childhood obesity are most likely to have long-term effects when they emphasize positive parenting practices. Parents' sensitivity and constructive scaffolding behaviors are related to children's self-regulation skills, which are robust predictors of healthy eating habits and body mass index (BMI). For example, children who have difficulty with self-regulation by age 3 have a higher BMI through age 12. Importantly, these relations may be causal: Adults who are taught self-regulation skills appear more successful in maintaining healthy eating habits over time. As a preventive intervention, Recipe 4 Success is implemented when children are 2, the point at which deliberate self-regulation skills are starting to emerge and develop rapidly and taste preferences are being formed. Recipe 4 Success is designed for families living in poverty because parents are less likely to provide sensitive scaffolding and children are less likely to display well-developed self-regulation skills and healthy eating habits under conditions of economic adversity. Finally, Recipe 4 Success was created to be integrated into Early Head Start to expedite wide-spread dissemination and easy sustainability and to enhance the efficacy of this nation-wide home visit program. If successful, this will be one of the first preventive interventions to improve either toddler's self-regulation skills or their healthy eating habits and BMI.

ELIGIBILITY:
Inclusion Criteria:

* Family lives in York, Allentown, Williamsport/Lock Haven Pennsylvania
* Family enrolled in Early Head Start home visit program
* Target child 18-36 months old at beginning of study

Exclusion Criteria:

* Family considered "in crisis" by home visitor (i.e., not able to focus on new intervention lessons because of child custody, family violence, mental health, or housing issues that currently demand parents' full attention)

Ages: 18 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2013-04-05 (Actual); Primary Completion 2014-02-27 (Actual); Study Completion 2014-02-27 (Actual)

PRIMARY OUTCOMES:
Change in percentage of healthy meals consumed | Change across three months, from baseline to post-intervention
  Daily food diaries were collected across three 24-hour periods. The percentage of meals that included at least one fruit and/or vegetable, at least one source of protein, and that did not include any sweets or junk food was calculated.
Change in willingness to eat healthy food | Change across three months, from baseline to post-intervention
  As part of the study assessment battery, parents were given novel healthy foods, such as dried seaweed, and asked to see if their children would like to eat them. The percentage of novel foods that children at least tasted was calculated.
Change in healthy body weight | Change across three months, from baseline to post-intervention
  Children's weight and height were collected with standardized scales and tape measures.
Change in children's self-control skills | Change across three months, from baseline to post-intervention
  Children completed a snack delay task in which an M&M was placed on a plate but the interviewer asked the children to wait 5-60 seconds before eating the M&M. The percentage of the four trials in which the child was able to wait the entire time requested before eating the M&M was calculated.
Change in children's attention | Change across three months, from baseline to post-intervention
  Children and their parents participated in three interaction tasks. Raters blind to study condition rated the ability of the children to concentrate and stay focused on what they were doing with their parents on a Likert scale with 1=almost never to 5 = almost always.
Change in children's compliance | Change across three months, from baseline to post-intervention
  Parents' completed the 8-item compliance subscale of the well-validated Infant and Toddler Social and Emotional Assessment. Each item was rated on a Likert scale with 1 = not true to 3 = very true.
Change in parents' sensitive scaffolding | Change across three months, from baseline to post-intervention
  Children and their parents participated in three interaction tasks. Raters blind to study condition rated the ability of the parents to sensitively scaffold their children's learning of a new task on a Likert scale with 1=almost never to 5 = almost always.
Change in parents' competent parenting | Change across three months, from baseline to post-intervention
  Children and their parents participated in three interaction tasks. Raters blind to study condition rated the overall competence of the parents on four items such as "The parent seemed very effective in interacting with the child" on a Likert scale with 1=almost never to 5 = almost always.
Change in parents' supportive feeding behaviors | Change across three months, from baseline to post-intervention
  As part of the study assessment battery, parents were given novel healthy foods, such as dried seaweed, and asked to see if their children would like to eat them. Interviewers blind to study condition rated whether or not parents engaged in four behaviors for each specific snack, such as "Parent modeled enjoyment of health food by tasting it her/himself." The percentage of times parents demonstrated such supportive feeding behaviors was calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Nix, Ph.D., Principal Investigator — University of Wisconsin-Madison (previously Pennsylvania State Univeristy)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nix RL, Francis LA, Feinberg ME, Gill S, Jones DE, Hostetler ML, Stifter CA. Improving Toddlers' Healthy Eating Habits and Self-regulation: A Randomized Controlled Trial. Pediatrics. 2021 Jan;147(1):e20193326. doi: 10.1542/peds.2019-3326. PMID 33372118